CLINICAL TRIAL: NCT07146646
Title: A Phase II Trial of Trifluridine/Tipiracil Plus Oxaliplatin in Patients With Advanced or Metastatic Biliary Tract Cancer Following First-Line Therapy
Brief Title: Trifluridine/Tipiracil + Oxaliplatin in Participants With Advanced or Metastatic Biliary Tract Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2225
Record Dates: First submitted 2025-08-12; First posted 2025-08-28 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Biliary Tract Cancer; Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Cancer; Gallbladder Carcinoma
Keywords: Trifluridine/tipiracil; FTD/TPI; Oxaliplatin
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms | interventions — trifluridine tipiracil drug combination; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FTD/TPI plus oxaliplatin (Experimental): Participants will complete 14-day treatment cycles of FTD/TPI plus oxaliplatin, continuing until disease progression, intolerable toxicities, or participant withdrawal from the trial.
  Interventions: Drug: Trifluridine/tipiracil; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Trifluridine/tipiracil — FTD/TPI will be taken by mouth on Days 1-5 of the 14-day treatment cycle. The starting does is 25mg/m2 twice per day.
  Other Names: FTD/TPI
Drug: Oxaliplatin — Oxaliplatin is given on Day 1 of each 14-day cycle. It is given intravenously (by IV) over 2 hours.

SUMMARY:
Participants are eligible for this study who were treated for advanced biliary tract cancer (BTC) but the treatment either did not make the cancer better or is no longer working. The treatment for patients whose advanced BTC either did not make the cancer better or is no longer working is a combination of chemotherapy drugs called FOLFOX which consists of fluorouracil and oxaliplatin. Studies have shown that other treatments may work better to treat advanced BTC. In this study, investigators want to see if treating patients with the drug combination of trifluridine/tipiracil (FTD/TPI) and another drug called oxaliplatin works better than FOLFOX for advanced BTC as second-line therapy. FTD/TPI are pills that are taken by mouth, whereas oxaliplatin is given intravenously (by IV).

DETAILED DESCRIPTION:
BTCs are difficult to treat. It is estimated that in the United States (US) approximately 15,000-20,000 people will be diagnosed with a BTC per year. In 2024, liver and intrahepatic bile duct cancers were the 5th leading cause of death from cancer among men and 7th among women in the US (1). Most people with BTCs have cancer that has spread or cannot be removed with surgery, so systemic treatments are the only option. However, the median survival after being diagnosed with an advanced BTC is still only 4.5 months, so it is important that we find better treatment options (2).

This study is evaluating the combination of a medicine called trifluridine/tipiracil (FTD/TPI) and a medicine called oxaliplatin in treating advanced BTCs. While FTD/TPI has been used to treat other types of cancer, it is not yet approved to treat BTCs, so it is experimental. On the other hand, oxaliplatin is a medicine that has been previously used to treat BTCs.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed biliary tract cancer (BTC) including cholangiocarcinoma and gallbladder carcinoma. Individuals with ampullary cancers will not be considered eligible. Cancer must be advanced stage or metastatic.
* Participants must have received only one line of systemic therapy for advanced or metastatic BTCs.
* Note: Individuals who have either progressed or are intolerant to the prior therapy can be included in this study.
* Age >18 years on day of signing informed consent. Because no dosing or adverse event data are currently available on the use of FTD/TPI in individuals ≤18 years of age, children are excluded from this study.
* Performance status: ECOG performance status of 0 or 1.
* At least one index lesion is measurable based on RECIST 1.1.
* Participants must have organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelet count ≥75,000/mcL
  * AST (SGOT) ≤ 2.5 X institutional upper limit of normal or ≤ 5 × ULN for participants with liver metastases
  * ALT (SGPT) ≤ 2.5 X institutional upper limit of normal or ≤ 5 × ULN for participants with liver metastases
  * Total bilirubin ≤ 1.5 × ULN or direct bilirubin ≤ ULN for participants with bilirubin levels >1.5 x ULN
  * Serum Creatinine ≤ 1.5 x upper limit of normal (ULN) or creatinine clearance ≥60 mL/min for participants with creatinine levels >1.5 x ULN (Cockcroft-Gault method)
* Participants must have recovered adequately from any major surgery, prior to starting therapy.
* Participants must have the ability to understand and the willingness to sign a written informed consent document.
* Agree to use adequate method of contraception.

Exclusion Criteria:

* Participants receiving any other investigational agents.
* Participant has received investigational therapy within 4 weeks or within 5 half-lives of the therapeutic agent (whichever is shorter).
* Received more than one line of systemic therapy for bile duct cancer. Adjuvant therapy will not be counted as line of systemic therapy.
* Receiving systemic steroid therapy (>10mg prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Prior treatment with FTD/TPI or oxaliplatin.
* Known additional malignancy that currently requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has already undergone potentially curative therapy.
* Known central nervous system metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are stable without evidence of new or enlarging brain metastases and are not using steroids for at least 7 days prior to trial treatment.
* Active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids (> 10 mg/day or equivalent of prednisone) or immunosuppressive agents. (thyroid disease and diabetes are allowed)
* Interstitial lung disease or active, non-infectious pneumonitis.
* Active infection requiring systemic antibiotics.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the individual's participation for the full duration of the trial, or is not in the best interest of the individual to participate, in the opinion of the treating investigator.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial, in the opinion of the treating investigator.
* Participants with uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations/substance abuse disorders that would limit compliance with study requirements.
* Participants pregnant or breastfeeding expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 5 months after the last dose of trial treatment. Pregnant or breastfeeding women are excluded from this study because it is unknown if the combination of FTD/TPI and oxaliplatin create the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study drug combination, breastfeeding should be discontinued if the mother is enrolled on this trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) by RECIST v1.1 | Every 8 weeks until treatment discontinuation, up to 6 months
  DCR is the percentage of participants whose cancer did not get worse after treatment (i.e. the percentage of participants who had CR, PR, or SD, as defined below), and this will be measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
  Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions. Partial Response (PR) is defined as a 30% decrease in the sum of diameters of target lesions. Progressive Disease (PD) is defined as a 20% increase in the sum of diameters of target lesions with an absolute increase of at least 5 millimeters (mm) or the appearance of one or more new lesions. Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.

SECONDARY OUTCOMES:
Safety and tolerability | Day 1
  Measured by the grade of adverse events (AEs) per CTCAE version 5.0
Safety and tolerability | At treatment discontinuation, up to 6 months
  Measured by the grade of adverse events (AEs) per CTCAE version 5.0
Safety and tolerability | 30 days post-study treatment discontinuation, up to 6 months
  Measured by the grade of adverse events (AEs) per CTCAE version 5.0
Safety and tolerability | Day 1
  Measured by the incidence of adverse events (AEs)
Safety and tolerability | At treatment discontinuation, up to 6 months
  Measured by the incidence of adverse events (AEs)
Safety and tolerability | 30 days post-study treatment discontinuation, up to 6 months
  Measured by the incidence of adverse events (AEs)
Safety and tolerability | Day 1
  Measured by the duration of adverse events (AEs)
Safety and tolerability | At treatment discontinuation, up to 6 months
  Measured by the duration of adverse events (AEs)
Safety and tolerability | 30 days post-study treatment discontinuation, up to 6 months
  Measured by the duration of adverse events (AEs)
Objective response rate (ORR) by RECIST v1.1 | Every 8 weeks until treatment discontinuation, up to 6 months
  ORR is the percentage of participants whose cancer got better after treatment (i.e. the percentage of participants who had CR or PR, as defined below), and this will be measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
  Per RECIST v1.1, Complete Response (CR) is defined as disappearance of all target lesions. Partial Response (PR) is defined as a 30% decrease in the sum of diameters of target lesions. Progressive Disease (PD) is defined as a 20% increase in the sum of diameters of target lesions with an absolute increase of at least 5 millimeters (mm) or the appearance of one or more new lesions. Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Progression free survival (PFS) | 2 years post-study treatment
  Progression-Free Survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Overall survival (OS) | 2 years post-study treatment
  Overall survival (OS) is defined as the duration of time from start of treatment to time of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Madison Conces, MD, Principal Investigator — Case Comprehensive Cancer Center, University Hospitals
Locations (2):
- United States (2):
  - University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 1 year after completion of the study
Access Criteria: Access available after completion of the study

REFERENCES:
- [Background] Siegel RL, Giaquinto AN, Jemal A. Cancer statistics, 2024. CA Cancer J Clin. 2024 Jan-Feb;74(1):12-49. doi: 10.3322/caac.21820. Epub 2024 Jan 17. PMID 38230766
- [Background] Nghiem V, Wood S, Ramachandran R, Williams G, Outlaw D, Paluri R, Kim YI, Gbolahan O. Short- and Long-Term Survival of Metastatic Biliary Tract Cancer in the United States From 2000 to 2018. Cancer Control. 2023 Jan-Dec;30:10732748231211764. doi: 10.1177/10732748231211764. PMID 37926828